CLINICAL TRIAL: NCT01573169
Title: PREvention of VENous Thromboembolism In Hemorrhagic Stroke Patients
Acronym: PREVENTIHS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial has been terminated prematurely after the randomization of 73 patients due to a lack of funding.
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Maurizio Paciaroni, Principal Investigator, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREVENTIHS
Record Dates: First submitted 2012-03-31; First posted 2012-04-06 (Estimated); Results first posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Hemorrhagic Stroke; Venous Thromboembolism; Deep Venous Thrombosis
Keywords: hemorrhagic stroke; venous thromboembolism; prevention
MeSH Terms: conditions — Hemorrhagic Stroke; Venous Thromboembolism; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low weight molecular heparin (Experimental): enoxaparin 0.4 ml subcutaneous per day
  Interventions: Drug: Enoxaparin
- standard therapy (Placebo Comparator): Graduated compression stockings and/or intermittent pneumatic compression and/or early mobilization
  Interventions: Other: Graduated compression stockings and/or intermittent pneumatic compression and/or early mobilization

INTERVENTIONS:
Drug: Enoxaparin — enoxaparin 0.4 ml sc per day for 10 days started 72 hours after the stroke
  Arms: low weight molecular heparin
Other: Graduated compression stockings and/or intermittent pneumatic compression and/or early mobilization — placebo standard therapy
  Arms: standard therapy

SUMMARY:
Patients with cerebral hemorrhage (ICH) have a high risk of venous thromboembolism. Intermittent pneumatic compression combined with elastic stockings have been shown to be superior to elastic stockings alone in reducing the rate of asymptomatic deep vein thrombosis after ICH in a randomized trial (4.7% vs. 15.9%). Graduated compression stockings alone are ineffective in preventing deep vein thrombosis in patients with ischemic or hemorrhagic stroke. Less clear is the role of anticoagulation in the prevention of venous thromboembolism in patients with ICH because the use of anticoagulants may cause an enlargement of the hematoma. In a multicenter, randomized trial, the investigators will assess the efficacy and safety of enoxaparin in the prevention of venous thromboembolism in patients with spontaneous intracerebral hemorrhage. Enoxaparin (40 mg once daily) or standard therapy (graduated compression stockings and/or intermittent pneumatic compression and/or early mobilization) will be given subcutaneously for not less than 10 days beginning after 72 hours from stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial spontaneous hemorrhage on brain CT scan
* Intracranial hemorrhage during treatment with oral anticoagulants
* Bedridden patients (item 6 of NIHSS: motor leg points 3 or 4 or severe ataxia for cerebellar hemorrhage).

Exclusion Criteria:

* cerebral hemorrhage due to intracranial vascular malformation
* rebleeding on CT scan after 72 hours from stroke (before randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-05; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Unit, Perugia, Italy

REFERENCES:
- [Background] Paciaroni M, Agnelli G, Venti M, Alberti A, Acciarresi M, Caso V. Efficacy and safety of anticoagulants in the prevention of venous thromboembolism in patients with acute cerebral hemorrhage: a meta-analysis of controlled studies. J Thromb Haemost. 2011 May;9(5):893-8. doi: 10.1111/j.1538-7836.2011.04241.x. PMID 21324058
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Paciaroni M, Agnelli G, Alberti A, Becattini C, Guercini F, Martini G, Tassi R, Marotta G, Venti M, Acciarresi M, Mosconi MG, Marcheselli S, Fratticci L, D'Amore C, Ageno W, Versino M, De Lodovici ML, Carimati F, Pezzini A, Padovani A, Corea F, Scoditti U, Denti L, Tassinari T, Silvestrelli G, Ciccone A, Caso V. PREvention of VENous Thromboembolism in Hemorrhagic Stroke Patients - PREVENTIHS Study: A Randomized Controlled Trial and a Systematic Review and Meta-Analysis. Eur Neurol. 2020;83(6):566-575. doi: 10.1159/000511574. Epub 2020 Nov 13. PMID 33190135

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No wash-out, nor run-in events.
Period: Overall Study
Arm/Group | Low Weight Molecular Heparin | Standard Therapy
Started | 38 | 35
Completed | 38 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Weight Molecular Heparin | Standard Therapy | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (13.7) | 71.5 (11.6) | 70.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 22 | 18 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Obesity [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic and Asymptomatic Venous Thromboembolism
Description: Symptomatic venous thromboembolism (deep venous thrombosis and/or pulmonary embolism) and asymptomatic deep venous thrombosis on ultrasound examination
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Weight Molecular Heparin | Standard Therapy
Number analyzed (Participants) | 38 | 35
Participants | 6 | 7

2. Secondary Outcome: Bleedings
Description: symptomatic and asymptomatic intra and extracranial bleedings
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Weight Molecular Heparin | Standard Therapy
Number analyzed (Participants) | 38 | 35
Participants | 1 | 3

3. Secondary Outcome: Mortality
Description: mortality of any cause
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Weight Molecular Heparin | Standard Therapy
Number analyzed (Participants) | 38 | 35
Participants | 7 | 6

4. Secondary Outcome: Disability
Description: modified Rankin Scale (mRS) equal to and greater than 3.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Weight Molecular Heparin | Standard Therapy
Number analyzed (Participants) | 38 | 35
Participants | 27 | 30

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Low Weight Molecular Heparin | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 7/38 | 6/35
Serious Adverse Events (participants affected / at risk) | 1/38 | 3/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Weight Molecular Heparin (N=38) | Standard Therapy (N=35)
extracranial bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intracranial bleedings (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT01573169/Prot_SAP_ICF_000.pdf